CLINICAL TRIAL: NCT00726648
Title: Double-blind, Placebo-controlled, Randomized, Parallel-group Study in Subjects With Relapsing Forms of Multiple Sclerosis to Evaluate the Effects of Different CDP323 Doses on Biomarker Patterns as Well as on Safety and Tolerability.
Brief Title: CDP323 Biomarker Study
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Collaborators: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: C32325; EudraCT 2008-000147-34; IND 74863
Record Dates: First submitted 2008-07-29; First posted 2008-08-01 (Estimated); Last update posted 2011-09-12 (Estimated); Status verified 2009-08

CONDITIONS: Relapsing Multiple Sclerosis
Keywords: CDP323; Relapsing multiple sclerosis; Blood biomarkers
MeSH Terms: interventions — CDP323

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- 1 (Experimental)
  Interventions: Drug: CDP323; Drug: Placebo
- 2 (Experimental)
  Interventions: Drug: CDP323; Drug: Placebo
- 3 (Experimental)
  Interventions: Drug: CDP323; Drug: Placebo
- 4 (Experimental)
  Interventions: Drug: CDP323; Drug: Placebo
- 5 (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CDP323 — 50mg capsules, 100mg bid for 4 weeks
  Arms: 2
Drug: CDP323 — 250mg capsules, 500mg bid for 4 weeks
  Arms: 3
Drug: CDP323 — 250mg capsules, 1000mg bid for 4 weeks
  Arms: 4
Drug: CDP323 — 250mg capsules, 1000mg daily for 4 weeks
  Arms: 1
Drug: Placebo — placebo capsules for 4 weeks

SUMMARY:
Comparison of the effects of different CDP323 doses given over a period of four weeks on blood biomarkers in subjects with relapsing forms of multiple sclerosis.

ELIGIBILITY:
Inclusion Criteria:

* Female and male subjects aged 18-65 years
* Relapsing form of MS with at least one clinical relapse in the 24 months before screening;
* Screening EDSS score of 0-6.5;
* Must be fully immunocompetent
* Female subjects of childbearing potential must agree to practice contraception methods

Exclusion Criteria:

* Any conditions that could interfere with the contrast-enhanced MRI;
* Any clinically significant disease state or findings other than MS;
* Any clinically significant deviation from the pre-defined ranges for laboratory tests;
* Concomitant treatment with MS disease modifying drugs

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2008-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamic parameters related to leukocyte trafficking | 4 weeks

SECONDARY OUTCOMES:
Standard and disease-related safety variables | 4 weeks
Class-related safety parameters | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — UCB Pharma
Locations (2):
- United Kingdom (2):
  - Tooting, London
  - Croydon, Surrey

REFERENCES:
- [Derived] Wolf C, Sidhu J, Otoul C, Morris DL, Cnops J, Taubel J, Bennett B. Pharmacodynamic consequences of administration of VLA-4 antagonist CDP323 to multiple sclerosis subjects: a randomized, double-blind phase 1/2 study. PLoS One. 2013;8(3):e58438. doi: 10.1371/journal.pone.0058438. Epub 2013 Mar 5. PMID 23472197